CLINICAL TRIAL: NCT05174325
Title: Phase II Exploratory Study of the Effectiveness of Neoadjuvant Chemotherapy Combined With PD-1 Monoclonal Antibody in the Treatment of Esophageal Squamous Cell Carcinoma: a Prospective, Single-center, Single-arm Study
Brief Title: Effectiveness of Neoadjuvant Chemotherapy Combined With PD-1 Monoclonal Antibody in the Treatment of Operable Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20211210
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — sintilimab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Pre-operative Sintilimab + chemotherapy
  Interventions: Drug: Sintilimab + chemotherapy

INTERVENTIONS:
Drug: Sintilimab + chemotherapy — Biological : Sintilimab 100mg: 10ml Method of administration: 200mg IV D1 Q3W. Drug: Cisplatin Injection Specification: 75mg/m2, IV D1 Q3W. Drug: Albumin Paclitaxel Injection specifications: 260mg/m2, IV D1 Q3W.

SUMMARY:
This study aims to evaluate the efficacy of sintilimab combined with concurrent chemotherapy as a neoadjuvant treatment for patients with operable esophageal squamous cell carcinoma. It will also evaluate the changes in the immune microenvironment of tumor specimens before and after the medication, and predict the operable period (stage I~III) Patients with thoracic esophageal squamous cell carcinoma were treated with neoadjuvant chemotherapy combined with PD-1 monoclonal antibody, and the effect of neoadjuvant chemotherapy combined with PD-1 monoclonal antibody was evaluated by detecting the changes of microbial diversity and metabolites in stool samples before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥18 years old and ≤75 years old; 2) Patients with stage I~III thoracic esophageal squamous cell carcinoma diagnosed by histopathological examination (excluding mixed adenosquamous carcinoma and other pathological types); 3) ECOG PS score is 0 or 1; 4) According to RECIST v1.1 version, there is at least one measurable lesion; 5) It has sufficient organ and bone marrow function, defined as follows: 6) Blood routine: absolute neutrophil count (ANC)≥1.5×109/L; platelet count (PLT)≥100×109/L; hemoglobin content (HGB)≥9.0 g/dL. Liver function: Patients without liver metastases require serum total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN. Renal function: creatinine clearance rate (Ccr) ≥60 mL/min (calculated by Cockcroft/Gault formula): female: Ccr= (140-years) x body weight (kg) x 0.85 72 x serum creatinine (mg/dL) male: Ccr= (140-years) x body weight (kg) x 1.00 72 x serum creatinine (mg/dL). Adequate coagulation function is defined as the international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; if the subject is receiving anticoagulation therapy, as long as the PT is within the proposed range of anticoagulation drugs; 7) Expected survival time ≥ 12 weeks; 8) Sign a written informed consent form and be able to comply with the visit and related procedures stipulated in the plan.

Exclusion Criteria:

* 1) Refuse to participate; 2) Patients with esophageal squamous cell carcinoma who are diagnosed as stage IV or have surgical contraindications or refuse surgery; 3) Patients who have a higher risk of bleeding or perforation due to the tumor's obvious invasion of the adjacent organs (aorta or trachea) of the esophageal lesion, or patients who have formed a fistula; 4) Have previously received anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibody therapy, or any other antibodies targeting T cell costimulation or checkpoint pathways as specific targets or drug; 5) Participate in another interventional clinical study at the same time, unless participating in an observational (non-interventional) clinical study or in the follow-up phase of an interventional study; 6) Have received systemic systemic treatment with anti-tumor indications Chinese herbal medicine or immunomodulatory drugs (including thymosin, interferon, interleukin, etc.) within 2 weeks before the first administration; 7) Have used immunosuppressive drugs within 1 week before enrollment, excluding nasal spray, inhalation or other local glucocorticoids or physiological doses of systemic glucocorticoids (ie no more than 10mg/day prednisone Or equivalent doses of other glucocorticoids), or use hormones to prevent allergy to contrast agents; 8) Receive live attenuated vaccine within 4 weeks before the first dose of study treatment or plan to receive the live attenuated vaccine during the study period; Note: It is allowed to receive the inactivated virus vaccine for seasonal influenza by injection within 4 weeks before the first dose; but it is not allowed to receive Live attenuated influenza vaccine; 9) Major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study treatment or expected major surgery during the study treatment period; 10) Prior to the first dose of study treatment, there was no recovery to the National Cancer Institute General Adverse Event Terminology version 5.0 (NCI CTCAE version 5.0) 0 or 1 toxicity (excluding hair loss, non-clinical) caused by previous anti-tumor therapy Significant and asymptomatic laboratory abnormalities); 11) Known active autoimmune disease and need symptomatic treatment or a history of the disease within the past 2 years (Vitiligo, psoriasis, hair loss or Grave's disease that does not require systemic treatment within the past 2 years, only need Patients with hypothyroidism under thyroid hormone replacement therapy and type I diabetes who only require insulin replacement therapy can be included in the group); 12) Known history of primary immunodeficiency; 13) Known to have active tuberculosis; 14) Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation; 15) Known to be allergic to any monoclonal antibody or chemotherapeutic drug (paclitaxel, cisplatin) preparations or excipient ingredients; 16) People with known HIV infection (HIV antibody positive); 17) Any arterial thromboembolic events, including myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack occurred within 6 months before being selected for treatment; 18) Significant malnutrition, such as intravenous supplementation of nutrient solutions; unless the malnutrition is corrected more than 4 weeks before the first dose of study treatment; 19) History of bowel obstruction or the following diseases: inflammatory bowel disease or extensive bowel resection (partial colectomy or extensive small bowel resection, complicated by chronic diarrhea), Crohn's disease, ulcerative colitis; 20) Known to have acute or chronic active hepatitis B (HBsAg positive and HBV DNA viral load ≥103 copies/mL or >200IU/ml) or acute or chronic active hepatitis C HCV antibody positive and HCV RNA Positive); 21) Suffer from interstitial lung disease that requires steroid therapy; 22) Female patients who are pregnant or breastfeeding; 23) Other acute or chronic diseases, mental illnesses, or abnormal laboratory test values that may cause the following results: increase the risk related to study participation or study drug administration, or interfere with the interpretation of the study results, and the patients shall be treated according to the judgment of the investigator Listed as not eligible to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete remission (PCR) | 4 weeks after surgery
  Primary tumor or lymph node surgery specimen pathological examination without residual tumor cell

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 4 weeks after surgery
  Objective Response Rate Determine the tumor shrinkage rate, tumor boundary and the adhesion of tumor
Radiographic response | From date of treatment allocation and during treatment period up to 3 months
  To assess radiographic response to neoadjuvant pembrolizumab with concurrent chemoradiotherapy using RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of soochow university, Suzhou, Jiangsu, China

REFERENCES:
- [Result] Huang B, Shi H, Gong X, Yu J, Xiao C, Zhou B, Liang Z, Li X. Comparison of efficacy and safety between pembrolizumab combined with chemotherapy and simple chemotherapy in neoadjuvant therapy for esophageal squamous cell carcinoma. J Gastrointest Oncol. 2021 Oct;12(5):2013-2021. doi: 10.21037/jgo-21-610. PMID 34790369
- [Result] Kudo T, Hamamoto Y, Kato K, Ura T, Kojima T, Tsushima T, Hironaka S, Hara H, Satoh T, Iwasa S, Muro K, Yasui H, Minashi K, Yamaguchi K, Ohtsu A, Doki Y, Kitagawa Y. Nivolumab treatment for oesophageal squamous-cell carcinoma: an open-label, multicentre, phase 2 trial. Lancet Oncol. 2017 May;18(5):631-639. doi: 10.1016/S1470-2045(17)30181-X. Epub 2017 Mar 15. PMID 28314688
- [Result] Kojima T, Shah MA, Muro K, Francois E, Adenis A, Hsu CH, Doi T, Moriwaki T, Kim SB, Lee SH, Bennouna J, Kato K, Shen L, Enzinger P, Qin SK, Ferreira P, Chen J, Girotto G, de la Fouchardiere C, Senellart H, Al-Rajabi R, Lordick F, Wang R, Suryawanshi S, Bhagia P, Kang SP, Metges JP; KEYNOTE-181 Investigators. Randomized Phase III KEYNOTE-181 Study of Pembrolizumab Versus Chemotherapy in Advanced Esophageal Cancer. J Clin Oncol. 2020 Dec 10;38(35):4138-4148. doi: 10.1200/JCO.20.01888. Epub 2020 Oct 7. PMID 33026938
- [Result] van den Ende T, de Clercq NC, van Berge Henegouwen MI, Gisbertz SS, Geijsen ED, Verhoeven RHA, Meijer SL, Schokker S, Dings MPG, Bergman JJGHM, Haj Mohammad N, Ruurda JP, van Hillegersberg R, Mook S, Nieuwdorp M, de Gruijl TD, Soeratram TTD, Ylstra B, van Grieken NCT, Bijlsma MF, Hulshof MCCM, van Laarhoven HWM. Neoadjuvant Chemoradiotherapy Combined with Atezolizumab for Resectable Esophageal Adenocarcinoma: A Single-arm Phase II Feasibility Trial (PERFECT). Clin Cancer Res. 2021 Jun 15;27(12):3351-3359. doi: 10.1158/1078-0432.CCR-20-4443. Epub 2021 Jan 27. PMID 33504550